CLINICAL TRIAL: NCT03749486
Title: To Assess if Using a High Resolution Immersion Ultrasound Measurement Improves Intraocular Lens Power Calculation
Brief Title: High Resolution Immersion Ultrasound for iIOL Power Calculation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ArcScan
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Cataract
Keywords: Cataract surgery; High resolution immersion ultrasound
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ArcScan (Experimental): High resolution immersion ultrasound measurement before Cataract surgery
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery — Cataract surgery will be done following ArcScan measurement

SUMMARY:
Assess is the additional use of high resolution immersion ultrasound measurements improve the refractive outcome after cataract surgery.

DETAILED DESCRIPTION:
Since the beginning of biometry, immersion ultrasound was shown to be accurate and reproducible. It is important to distinguish between immersion ultrasound techniques and contact ultrasound. The later was shown to be less accurate and examiner dependent.

Although immersion ultrasound has been improved significantly and novel high resolution ultrasound devices are available, the drawback of this technique is that measurement s take longer compared to optical biometry. The advantage of immersion ultrasound is that structures behind the iris are visible, whereas in optical biometry only structures within the pupil are visible.

Immersion ultrasound as well optical biometry can be used to calculate the needed power of an intraocular lens (IOL) to achieve the aimed post-operative refraction. Although IOL power calculation improved within the last decades, refractive surprises occur, especially in cases with very short eyes.

The estimation of the post-operative IOL position and therefore the estimated anterior chamber depth (ACD) is presently the main source of error (35% to 42%) in IOL power calculation and therefore for the refractive outcome of the patients after cataract surgery. Early IOL power calculation formulae, such as the Binkhorst I formula, used a fixed ACD value to predict the position of the IOL, but the refractive results were not appropriate because the post-operative position of the IOL varied significantly between patients. Later observations showed a correlation between the axial eye length and the post-operative ACD (more myopic eyes showed a larger ACD post-operatively). These correlations were taken into account in later developed formulas (such as the Binkhorst II formula). Olsen et al. measured the post-operative ACD and substituted the predicted post-operative ACD with the true, post-operative ACD in each case. The result after correcting the IOL position was a highly accurate IOL power calculation, where no fudge factors were needed. Presently the pre-operatively measured ACD is taken into account for several IOL power calculation formulas, such as the Haigis formula, the Holladay II formula and the Olsen formula. However, this new generation of formulas use the pre-operative ACD, without considering the thickness of the crystalline lens. The ACD is measured as the distance between the anterior surface of the cornea (anatomically speaking this should be the posterior surface of the cornea, but in an optical context, as in IOL power calculations, the anterior surface is used) and the anterior surface of the crystalline lens . Therefore the thickness of the crystalline lens has a significant impact on the predicted post-operative position of the IOL. This parameter was first taken into account by Olsen and later modified by Norrby.

It should be mentioned that IOL power calculations developed from theoretical calculations based on Gaussian optics to regression formulas, such as the SRK formula that uses retrospective data of a large number of patients. All these findings suggest that proper measurements not only of the dimensions of the crystalline lens but also of the lens capsule after removing the crystalline lens are necessary to improve IOL power calculation.

A prototype of a combination of an anterior segment OCT (VISANTE; Carl Zeiss Meditec AG) and an operating microscope (OPMI 200; Carl Zeiss Meditec AG) was introduced that allowed measurements of the crystalline lens as well as the lens capsule itself after removing the crystalline lens of cataract patients intraoperatively. This device uses OCT technology to create high resolution B-scans (=images) of the anterior segment of the eye. The OCT was shown to be highly reproducible for ACD measurements pre-operatively and small changes of the IOL/crystalline lens can be detected.

This prototype set-up was used in a previous study published in the journal "Investigative Ophthalmology & Visual Science". It was shown that intra-operative measurements of the anterior lens capsule were a better predictor for the post-operative lens position than other factors and could improve the refractive outcome theoretically. Furthermore it was shown that intra-operatively measured anterior chamber depth is useful to predict refractive outcome using fourth-generation formulae. A further study aimed to observe, whether the postoperative refractive outcome could be improved theoretically by using both pre- and intra-operative measurements for retrospective IOL power calculation with new eye models.

In a recent study a high resolution swept-source OCT was used to perform the measurements and results were very promising (DIATHLAS; Carl Zeiss Meditec AG, Germany).

However, disadvantage of swept-source OCT technology is that the measured area is only within the pupil, but structures behind the iris cannot be visualised.

Most recent findings suggest that measuring the equator of the lens capsule and the cilliary body could improve IOL power calculation.

One CE marked device that allows measurements behind the iris is the ArcScan Insight 100 scanner. This immersion ultrasound device is a precision high frequency device for imaging and biometry of the eye. A 20-60 MHz transducer scans the eye although its curvature approximates the anterior ocular surface. During this process the device produces images with 1 micron resolution of the cornea or the anterior segment. In addition, measurements can also be made of the anatomic structures comprising the anterior of the eye such as anterior chamber depth, angle-to-angle width, and sulcus-to-sulcus width, and pathologic structures, such as solid masses and cysts.

ELIGIBILITY:
Inclusion Criteria:

* Cataract
* Age 21 and older
* Able to understand the patient information
* Willing to follow the instructions and attend all follow-up visits
* Willing to sign informed consent prior to surgery

Exclusion Criteria:

* Relevant other ophthalmic diseases that are likely to reduce the refractive outcome, such as pseudoexfoliation syndrome, traumatic cataract, severe corneal scars
* Previous ocular surgeries on the study eye
* Patients who are not able to cooperate, with eccentric fixation or insufficient ability to fixate (tremor, nystagmus)
* Pregnant or lactating women (pregnancy testing will be performed preoperatively on women of reproductive age)

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Difference in mean absolute error in refractive outcome | 12 months
  The difference in refractive error will be measured using auto- and subjective refraction

SECONDARY OUTCOMES:
Anterior chamber depth and lens thickness measurement | 12 months
  Anterior chamber depth and lens thickness will be measured using the IOL Master 700
IOL tilt and decentration | 12 months
  IOL tilt and decentration will be assessed using the Purkinjemeter

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided